CLINICAL TRIAL: NCT05463510
Title: Dermoscopic Monitoring of Pediatric Melanocytic Nevi Regarding Pattern and Diameter Changes
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Esra Koku Aksu, Head of the Dermatology Department, MD, Istanbul Training and Research Hospital
Other Study IDs: Karar no:108 25.03.2022
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Nevus, Pigmented
MeSH Terms: conditions — Nevus, Pigmented

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric melanocytic nevus: 50 patients and 301 pediatric nevi were evaluated
  Interventions: Diagnostic Test: Videodermoscopy

INTERVENTIONS:
Diagnostic Test: Videodermoscopy — Patients who had records for at least twice with videodermoscopy every 3 months were included.

SUMMARY:
Childhood and adolescence are a dynamic process in terms of nevogenesis, and the development and growth of new melanocytic nevus is frequently observed. Melanomas, although rare, can also be seen in the pediatric age group. Therefore, nevus monitoring with videodermoscopy may be necessary in the pediatric age group. Aim of our study is to show the dynamic pattern and diameter modifications in pediatric nevi.

DETAILED DESCRIPTION:
Aim of our study is to show the dynamic pattern and diameter modifications in pediatric nevi. Patients who applied to the Dermatology Clinic of Istanbul Training and Research Hospital between January 2008 and January 2022, were diagnosed with pediatric melanocytic nevus clinically and dermoscopically were included. Patients who had records for at least twice with videodermoscopy every 3 months were included. In the study, 301 pediatric melanocytic nevi belonging to 50 patients were evaluated.

The following characteristics were recorded in a database specifically designed for the study:Demographic findings of the patients, nevus localization, nevus pattern (baseline and follow-up), nevus diameter (base line and follow-up at 3/12/36th months), histopathological results of nevi that underwent total excision were recorded. The change in nevus diameter during follow-up was measured in millimeters based on the longest axis. Presence of peripheral globules, outcome of peripheral globules, characteristics of peripheral globules were recorded. Characteristics of peripheral globules were evaluated according to being around the entire lesion (circumferential) versus focally presence, typical (uniform shape and colors) and being regular (single rim of globules or multiple rim of globules)

ELIGIBILITY:
Inclusion Criteria:

* Subjects <18 years of age
* Subjects who have dermoscopic diagnosis of melanocytic nevus
* Subjects who had dermoscopic follow up for at least 3 months

Exclusion Criteria:

* Subjects >18 years of age

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients who applied to the Dermatology Clinic of Istanbul Training and Research Hospital between January 2008 and January 2022, were diagnosed with pediatric melanocytic nevus clinically and dermoscopically were included. Patients who had records for at least twice with videodermoscopy every 3 months were included. In the study, 301 pediatric melanocytic nevi belonging to 50 patients were evaluated.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Pediatric nevi diameter change in millimeters | 3-36 months
  1.Nevus diameter change at 3/12/36th months (measurement of longest axis of nevus as millimeters with videodermoscopy)
Pediatric nevi pattern change | 3-36 months
  Nevus pattern change at 3/12/36th months (pattern is categorized as globular/reticular/homogenous/fibrillar/parallel furrow or combinations)
Presence of peripheral globules | 3-36 months
  Peripheral globules will be recorded if present and will be categorized as (increased, decreased or no change) at the 3/12/36th months

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Esra Koku Aksu, MD, Principal Investigator — Istanbul Teaching and Research Hospital
Locations (1):
- Istanbul Teaching and Research Hospital, Istanbul, Istanbul/Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Piazza CD, Yamada S, Marcassi AP, Maciel MG, Seize MP, Cestari SCP. Dermoscopic patterns of melanocytic nevi in children and adolescents: a cross-sectional study. An Bras Dermatol. 2017 May-Jun;92(3):340-344. doi: 10.1590/abd1806-4841.20175209. PMID 29186245
- [Result] Zalaudek I, Schmid K, Marghoob AA, Scope A, Manzo M, Moscarella E, Malvehy J, Puig S, Pellacani G, Thomas L, Catricala C, Argenziano G. Frequency of dermoscopic nevus subtypes by age and body site: a cross-sectional study. Arch Dermatol. 2011 Jun;147(6):663-70. doi: 10.1001/archdermatol.2011.149. PMID 21690528
- [Result] Fortina AB, Zattra E, Bernardini B, Alaibac M, Peserico A. Dermoscopic changes in melanocytic naevi in children during digital follow-up. Acta Derm Venereol. 2012 Jul;92(4):427-9. doi: 10.2340/00015555-1306. PMID 22367216